CLINICAL TRIAL: NCT05125705
Title: Treatment of Lateral Epicondylitis With Platelet-Rich Plasma Versus Saline: A Double-Blinded Randomized Placebo-Controlled Trial
Brief Title: PRP Versus Saline in Lateral Epicondylitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Kenon Chua Ser, Orthopaedic Surgery Registrar, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIRB1
Record Dates: First submitted 2021-10-23; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Lateral Epicondylitis, Unspecified Elbow
Keywords: platelet rich plasma; saline; randomised controlled trial
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the patients and the outcome assessor will be blinded in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma injection (Experimental): Patients will be treated with a single PRP injection, where 8 mL of whole blood will be collected and 2.5 mL of PRP will be given to the patient. Routine physiotherapy regimens will be implemented, similar to placebo arm.
  Interventions: Biological: Platelet rich plasma injection
- Saline injection (Placebo Comparator): Patients will be treated with 2.5 mL saline 0.9%. Routine physiotherapy regimens will be implemented, similar to intervention arm.
  Interventions: Other: Saline injection

INTERVENTIONS:
Biological: Platelet rich plasma injection — The PRP is prepared by RegenLab's RegenKit-THT, in accordance with operating instructions supplied with the kit. The device allows automated blood collection (8 mL) and blood component separation in closed circuit. After centrifugation at room temperature for 9 minutes at centrifugal force of 1500g, the RegenTHT tube is then inverted several times before re-suspension, allowing 4mL of PRP to be obtained for each tube. 2.5mL will be injected into patients
  Other Names: PRP
  Arms: Platelet rich plasma injection
Other: Saline injection — Saline injection
  Arms: Saline injection

SUMMARY:
Lateral epicondylitis (LE), also known as tennis elbow, has an estimated prevalence in the general population of 1% to 3%, peaking at age 45 years to 54 years and affect both men and women equally. A randomised controlled trial published in The Lancet showed that 83% of the patients suffering from LE of more than 6 weeks duration on wait-and-see policy recovered only after 1 year without any therapeutic interventions. The costs associated with LE is substantial as patients not only incur hefty healthcare costs but also lose their productivity owing to their long recovery period.

Currently, there is a paucity of evidence worldwide for the efficacy of PRP injections compared to control in LE. This randomised controlled trial aims to compare the efficacy of PRP versus placebo (saline) injections in adults with LE.

DETAILED DESCRIPTION:
The pathogenesis of LE was initially believed to be a generalised inflammatory process. However, in 1979, the pathology was better understood as invading immature fibroblasts disorganizing the normal collagen architecture of the elbow, associated with immature vascular responses to cellular repair. There is a variety of treatment modalities available for LE, varying from watchful waiting without any therapeutic interventions, pharmaceutical methods such as prescribing non-steroidal anti-inflammatory drugs, physiotherapy such as encouraging bracing and exercise, injections, and surgical modalities once non-surgical options fail.

For many years, injection with glucocorticoids has remained the mainstay of treatment. However, several studies have proven that the effects of corticosteroid injections do not seem to last in the long-term, amongst which a trial published in The Lancet showed that long-term differences at 52 weeks between injections and physiotherapy was significantly in favour of physiotherapy. Recently, many studies worldwide have demonstrated that platelet-rich-plasma (PRP) stimulates cartilage repair by actively secreting growth factors which activate cell proliferation and differentiation thereby promoting tissue regeneration. It has been postulated that PRP stimulates repair mechanisms within tendons and hence promote tendon healing.

However, there is a paucity of evidence worldwide for the efficacy of PRP injections compared to control in LE. Currently, PRP treatment is not formally recognized as a treatment modality for LE in Singapore, with the accepted indications for PRP treatment being limited to non-surgical treatment of acute muscle and ligamentous injuries, and the biological augmentation of acute Achilles tendon repairs.

This randomised controlled trial aims to compare the efficacy of PRP versus placebo (saline) injections in adults with LE.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age >21 years old
* History of chronic pain on the lateral side of the elbow and pain on lateral epicondyle on direct palpation and resisted dorsiflexion of the wrist for more than 3 months
* Ability of patients to provide informed consent

Exclusion Criteria:

* Previous tennis elbow surgery to affected elbow
* Previous corticosteroid injections to affected elbow
* Concurrent complementary and alternative medicine (CAM) treatments e.g. acupuncture
* Inflammatory diseases / infection / fracture / trauma
* Neck pain on ipsilateral side
* Chronic pain syndromes
* Malignancies
* Pregnant or lactating females
* Consistent use of NSAIDs within 48 hours of procedure
* Systemic use of corticosteroids within 2 weeks
* History of anemia, any blood disorders, hypothyroidism

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Patient-Related Tennis Elbow Evaluation (PRTEE) pain in affected arm | baseline
  Rates pain from 0 (no pain) to 10 (worst imaginable) for at rest, doing task with repeated arm movement, carrying plastic bag of groceries, when pain was least, when pain was worst
Patient-Related Tennis Elbow Evaluation (PRTEE) pain in affected arm | 6 weeks
  Rates pain from 0 (no pain) to 10 (worst imaginable) for at rest, doing task with repeated arm movement, carrying plastic bag of groceries, when pain was least, when pain was worst
Patient-Related Tennis Elbow Evaluation (PRTEE) pain in affected arm | 3 months
  Rates pain from 0 (no pain) to 10 (worst imaginable) for at rest, doing task with repeated arm movement, carrying plastic bag of groceries, when pain was least, when pain was worst
Patient-Related Tennis Elbow Evaluation (PRTEE) pain in affected arm | 6 months
  Rates pain from 0 (no pain) to 10 (worst imaginable) for at rest, doing task with repeated arm movement, carrying plastic bag of groceries, when pain was least, when pain was worst
Patient-Related Tennis Elbow Evaluation (PRTEE) functional disability | baseline
  Rates from 0 (no difficulty) to 10 (unable to do) on specific activities and usual activities. Specific activities include turning doorknob or key, carrying grocery bag or briefcase by handle, lifting full coffee cup or glass of milk to mouth, opening jars, pulling up pants, wringing out washcloths or wet towels. Usual activities include personal activities (dressing, washing), household work (cleaning, maintenance), work (job), recreational or sporting activities.
Patient-Related Tennis Elbow Evaluation (PRTEE) functional disability | 6 weeks
  Rates from 0 (no difficulty) to 10 (unable to do) on specific activities and usual activities. Specific activities include turning doorknob or key, carrying grocery bag or briefcase by handle, lifting full coffee cup or glass of milk to mouth, opening jars, pulling up pants, wringing out washcloths or wet towels. Usual activities include personal activities (dressing, washing), household work (cleaning, maintenance), work (job), recreational or sporting activities.
Patient-Related Tennis Elbow Evaluation (PRTEE) functional disability | 3 months
  Rates from 0 (no difficulty) to 10 (unable to do) on specific activities and usual activities. Specific activities include turning doorknob or key, carrying grocery bag or briefcase by handle, lifting full coffee cup or glass of milk to mouth, opening jars, pulling up pants, wringing out washcloths or wet towels. Usual activities include personal activities (dressing, washing), household work (cleaning, maintenance), work (job), recreational or sporting activities.
Patient-Related Tennis Elbow Evaluation (PRTEE) functional disability | 6 months
  Rates from 0 (no difficulty) to 10 (unable to do) on specific activities and usual activities. Specific activities include turning doorknob or key, carrying grocery bag or briefcase by handle, lifting full coffee cup or glass of milk to mouth, opening jars, pulling up pants, wringing out washcloths or wet towels. Usual activities include personal activities (dressing, washing), household work (cleaning, maintenance), work (job), recreational or sporting activities.
Visual analog scale (VAS) pain with resisted wrist extension | baseline
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with resisted wrist extension | 6 weeks
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with resisted wrist extension | 3 months
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with resisted wrist extension | 6 months
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with contraction of extensor carpi radialis brevis and extensor digitorum communis | baseline
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with contraction of extensor carpi radialis brevis and extensor digitorum communis | 6 weeks
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with contraction of extensor carpi radialis brevis and extensor digitorum communis | 3 months
  Rated from 0 (no pain) to 5 (extremely pain)
Visual analog scale (VAS) pain with contraction of extensor carpi radialis brevis and extensor digitorum communis | 6 months
  Rated from 0 (no pain) to 5 (extremely pain)
Ultrasound tendon | baseline
  Ultrasonographic changes in tendon thickness and color Doppler activity will be recorded
Ultrasound tendon | 6 months
  Ultrasonographic changes in tendon thickness and color Doppler activity will be recorded

IPD SHARING:
Plan to Share IPD: No